CLINICAL TRIAL: NCT07351695
Title: Assessment of Nutritional Status in Children With Cerebral Palsy
Brief Title: Assessment of Nutritional Status Using Mid-Upper Arm Circumference Z-Score in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Hülya Kayılıoğlu, Faculty Member, Muğla Sıtkı Koçman University
Other Study IDs: CP-220086
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Malnutrition in Children
Keywords: Cerebral palsy; Child nutrition disorders; Anthropometry; Body Mass Index; Feeding and Eating Disorders; Malnutrition; Motor Activity; Nutritional Status
MeSH Terms: conditions — Cerebral Palsy; Child Nutrition Disorders; Feeding and Eating Disorders; Malnutrition; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral Palsy: This observational study includes a single cohort of pediatric patients with a confirmed diagnosis of cerebral palsy. Participants are enrolled during routine outpatient follow-up visits at a tertiary care center.
  Within the cohort, participants are categorized according to nutritional status based on predefined anthropometric criteria and according to functional severity using established classification systems. No separate control group is included. Comparisons are performed within the cohort across nutritional status categories and functional severity levels to evaluate distributions and associations.

SUMMARY:
Children with cerebral palsy are at increased risk of malnutrition due to motor impairment, feeding difficulties, and chronic health problems. Accurate assessment of nutritional status in this population can be challenging, particularly when standard anthropometric measurements are difficult to obtain.

This observational study aims to evaluate nutritional status in children with cerebral palsy using the mid-upper arm circumference Z-score (MUACZ) and to examine its relationship with functional severity levels. Anthropometric measurements and clinical data will be collected during routine outpatient visits. Nutritional status will be classified using predefined reference standards, and associations with motor and feeding function classifications will be analyzed.

The findings of this study are expected to contribute to a better understanding of practical approaches for nutritional assessment in children with cerebral palsy across different ages and functional levels.

DETAILED DESCRIPTION:
Cerebral palsy is a non-progressive neurodevelopmental condition frequently associated with motor dysfunction, feeding difficulties, and impaired growth. Malnutrition remains a common and clinically important comorbidity in children with cerebral palsy and is associated with adverse health outcomes, including increased susceptibility to infections, reduced muscle strength, and diminished quality of life. Despite its clinical relevance, accurate nutritional assessment in this population is often complicated by postural limitations, contractures, and difficulties in obtaining reliable weight and height measurements.

This cross-sectional, observational study is designed to assess nutritional status in children with cerebral palsy using anthropometric indicators, with a particular focus on the mid-upper arm circumference Z-score (MUACZ). MUACZ is derived from age- and sex-adjusted reference standards and can be obtained with minimal equipment, making it potentially suitable for use across a wide range of functional severity levels.

The study will include pediatric patients with a confirmed diagnosis of cerebral palsy who attend routine follow-up visits at a tertiary care center. Anthropometric measurements, including mid-upper arm circumference, body mass index-for-age, and height-for-age Z-scores, will be recorded according to standardized procedures. Functional severity will be classified using the Gross Motor Function Classification System (GMFCS) and the Eating and Drinking Ability Classification System (EDACS).

Nutritional status will be categorized based on predefined Z-score thresholds. Statistical analyses will examine the distribution of nutritional status across functional severity levels and evaluate the performance of MUACZ in identifying undernutrition using established cutoff values. All analyses will be conducted using appropriate statistical software, and the study will adhere to relevant ethical standards, with informed consent obtained from parents or legal guardians.

This study does not involve any intervention or alteration of standard clinical care. Data are collected solely for observational and analytical purposes.

ELIGIBILITY:
Inclusion Criteria

* Children and adolescents with a confirmed diagnosis of cerebral palsy
* Age between 18 months and 18 years at the time of assessment
* Attendance at routine outpatient follow-up at the study center during the study period
* Availability of anthropometric measurements required for nutritional assessment
* Availability of functional classification using the Gross Motor Function Classification System (GMFCS) and/or the Eating and Drinking Ability Classification System (EDACS)
* Written informed consent obtained from a parent or legal guardian

Exclusion Criteria

* Presence of acute illness or infection at the time of assessment that could interfere with anthropometric measurements
* Known genetic syndromes or metabolic disorders affecting growth independently of cerebral palsy
* Incomplete clinical or anthropometric data preventing classification of nutritional status
* Previous major surgery or hospitalization within a period that could significantly influence nutritional measurements (as determined by the treating clinician)

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children and adolescents with a confirmed diagnosis of cerebral palsy who are followed at a tertiary referral center. Participants are recruited during routine outpatient follow-up visits and represent a wide spectrum of motor and feeding functional severity.
  The population includes patients across all levels of gross motor function and eating and drinking ability, allowing evaluation of nutritional status across varying degrees of functional impairment. Anthropometric and clinical data are collected as part of standard care, without any modification to routine clinical management.
  This population reflects a real-world clinical setting in which nutritional assessment is routinely performed in children with cerebral palsy, including those with severe motor and feeding limitations.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of undernutrition in children with cerebral palsy | At study enrollment (single assessment during routine outpatient visit).
  Undernutrition status will be determined using predefined anthropometric Z-score criteria. Undernutrition is defined as the presence of wasting (body mass index-for-age Z-score ≤ -2) and/or stunting (height-for-age Z-score ≤ -2), based on standardized growth references.

SECONDARY OUTCOMES:
Distribution of nutritional status across functional severity levels | At study enrollment.
  The distribution of undernutrition will be evaluated across functional severity categories as defined by the Gross Motor Function Classification System (GMFCS) and the Eating and Drinking Ability Classification System (EDACS).
Association between MUACZ and functional severity classifications | At study enrollment.
  The relationship between mid-upper arm circumference Z-score (MUACZ) values and functional severity levels (GMFCS and EDACS) will be analyzed using appropriate statistical methods.
Performance of MUACZ in identifying undernutrition | At study enrollment.
  The ability of MUACZ to identify undernutrition will be evaluated using receiver operating characteristic analysis with a predefined cutoff value (≤ -2).

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman Research and Training Hospital, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this study, including demographic variables, anthropometric measurements, and functional classification data.
Supporting Information: Analytic Code
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years following publication.
Access Criteria: Individual participant data will be made available to qualified researchers upon reasonable request. Requests will be reviewed by the corresponding author and require approval from the relevant institutional and/or ethics committees, where applicable. Data will be shared in de-identified form to protect participant privacy, and access may require a data use agreement specifying the intended use of the data.